CLINICAL TRIAL: NCT01290016
Title: MY LIFE Study - McGill Youth Lifestyle Intervention With Food and Exercise Study
Brief Title: Youth Lifestyle Intervention With Food and Exercise
Acronym: MYLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HW-10-03
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Healthy; Obesity
Keywords: randomized controlled trial; children; obesity; nutrition; exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control 6-8 yrs (Active Comparator): The group will receive information during the study about diet and exercise but will not receive the intervention till the end of the study protocol.
  Interventions: Behavioral: Control
- 2 servings dairy + exercise 6-8 yrs (Experimental): Subjects in this group will receive family based counseling to maintain the intake of 2 servings of dairy per day and also receive instruction on how to improve their physical activity.
  Interventions: Behavioral: 2 servings dairy + exercise
- 4 servings dairy + exercise 6-8 yrs (Experimental): Subjects in this group will receive family based counselling to maintain the intake of 4 servings of dairy per day and also receive instruction on how to improve their physical activity.
  Interventions: Behavioral: 4 servings dairy + exercise
- 4 servings dairy + exercise 9-12 yrs (Experimental): Subjects in this group will receive family based counselling to maintain the standard recommended intake of 4 servings of dairy per day for 9-14 year olds according to the Canada's Food Guide and also receive instruction on how to improve their physical activity.
  Interventions: Behavioral: 4 servings dairy + exercise
- Control 9-12 yrs (Active Comparator): The group will receive information during the study about diet and exercise but will not receive the intervention until 6 months into the study protocol.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: 2 servings dairy + exercise — Subjects in this group will receive family based counseling to maintain the intake of 2 servings of dairy per day and also receive instruction on how to improve their physical activity.
  Other Names: 2 servings of dairy and exercise
  Arms: 2 servings dairy + exercise 6-8 yrs
Behavioral: 4 servings dairy + exercise — Subjects in this group will receive family based counseling to increase intake of dairy to 4 servings per day and also receive instruction on how to improve their physical activity.
  Other Names: 4 servings of dairy and exercise
  Arms: 4 servings dairy + exercise 6-8 yrs; 4 servings dairy + exercise 9-12 yrs
Behavioral: Control — The group will receive information during the study about diet and exercise but will not receive the intervention until 6 months into the study protocol.
  Arms: Control 6-8 yrs; Control 9-12 yrs

SUMMARY:
Children who are overweight or obese can develop many health complications including diabetes, high blood pressure, high cholesterol and they break their bones more often than children who are of healthy body weights. Recent short-term studies in children suggest that increasing milk intake for 16 weeks begins to improve body composition and also reduces risk of developing diabetes. However, no study has been long enough to truly test for the benefits of high milk consumption on these conditions including bone. Both dietary and activity approaches to reducing obesity in children are suggested by health professionals and when combined are called lifestyle interventions. Therefore, McGill University has designed a 1-year intervention study focused on lifestyle improvements to reduce obesity in children 6 to 12 years of age. A control group will be monitored for the year, while two other groups will receive lifestyle interventions with standard recommended (2 servings a day) and high (4 servings a day) intakes of milk. The intervention will include 6 planning sessions to increase intakes of vegetables, fruits and milks along with more activity and less time watching television or using computerized games. Children will have muscle and fat measured using an x-ray device that also measures bone at the beginning, middle and end of the study. They will also have a small blood sample taken every 3 months to measure blood sugar, cholesterol and some nutrients. Changes over the study will demonstrate the benefits of lifestyle and milk interventions.

DETAILED DESCRIPTION:
Rationale: Childhood obesity is an increasingly major health care problem in Canada. Not only are approximately 30% of Canadian children overweight/obese, but they are developing significant sequelae including insulin resistance, hyperinsulinemia, hyperlipidemia, hypertension, and diabetes mellitus. Additionally obese children have lower bone mass, lower 25(OH)D concentrations and fracture more frequently. Canadian children on average do not meet the recommended intakes for vegetables and fruit and only half of those < 8 years old meet the recommended intakes for milk. Obese children are more likely to be inactive and spend more screen-time during their free time. There is promising childhood evidence that diets with 3 to 4 servings of milk support healthier body composition (lean mass and height) and improved insulin sensitivity in the short term and bone mass in the longer term. Family based interventions are effective in weight reduction in children. To date, a combined assessment of the benefits of improved intakes of milk plus active lifestyles in obese children on body composition, bone and blood biochemistry in a family intervention is lacking.

Objectives and Hypotheses:

1. To determine if a 1-year lifestyle intervention with planning sessions designed to improve diet and activity within the context of the family environment will reduce adiposity and elevate lean mass while supporting bone mass in obese children compared to a control group and if augmented intake of milk to 4 daily servings will result in superior changes. The primary outcome will be change in body mass index (BMI) Z-score along with waist circumference for assessment of adiposity; selected for ease of use in larger studies or clinics where body composition assessment is not feasible.

   Hypothesis: the lifestyle intervention will yield modest changes to adiposity and lean mass accompanied by no reductions in bone mass, but that the augmented milk intervention will yield superior reductions in adiposity and elevations in lean and bone mass and height growth. It is hypothesized that bone mass will be low and that maintenance of bone mass in the standard intervention will thereby be judged as inadequate.
2. To explain the hypothesized benefits of these interventions on lean, adipose and bone masses by measuring indicators of glucose metabolism, satiety and related gut hormones along with novel biomarkers of skeletal metabolism including osteocalcin, adiponectin and vitamin D.

   Hypothesis: high milk intake will associate with lower glucose, insulin, ghrelin and 1,25(OH)2D accompanied by higher 25(OH)D, osteocalcin, peptide YY and glucagon-like peptide 1.
3. Test if the intervention with higher milk servings is linked to changes in child eating behavior and satiety using the Child Eating Behavior Questionnaire to reflect eating in the child's normal environment.

Hypothesis: children randomized to the high milk intervention group will demonstrate improved scores on the satiety responsiveness component of the survey.

METHODS - Randomized Controlled Trial Ethics: This study was approved by the McGill University Institutional Review Board of the Faculty of Medicine in October 2010 and will also be conducted in compliance with the Tri-Council Policy Statement 2005 and in compliance with local regulation and laws governing research involving human subjects. Otherwise healthy obese children (6 to 12 years of age) will be recruited following informed consent. Upon completion, the control group will be offered the counseling (5 visits) intervention adjusted for age (i.e. counseling + basic anthropometric measurements only).

Population and Recruitment: Obese children (n=150) from West-Island Montreal and surrounding off island areas within 50 km of the Macdonald Campus of McGill University. Our approach to recruitment is to use mailings through Canada Post. This service is excellent and the result is that for a particular area (predominantly West Island Montreal and off island areas towards Ottawa) each household receives a brochure on the study inviting them to attend if they have a child who has a body mass index (BMI) in our range. A graph will be provided to guide the parents and they will be invited to call us for more information. Obesity will be defined on the basis of body mass index > 95th percentile for age according to the World Health Organization. In total 150 children 6 to 12 years of age will be recruited over a 6-month window. Those meeting entrance criteria will be randomized into 3 groups:

1. a control group with information only (counseling after 12 months for 6-8 year olds and after 6 months for 9-12 year olds);
2. a lifestyle intervention (planning/counseling to improve diet and activity)(6-8 year olds only);
3. the same lifestyle intervention augmented with a total of 4 servings of milk/milk products daily (6-12 year olds).

Study Protocol: Participants will be screened for entrance criteria at a visit 2 weeks prior to beginning the 1-year program. Upon confirmation of meeting inclusion criteria, families will be telephoned to confirm participation and then 6-8 year olds will be randomized into the 3 groups stratified for sex and the 9-12 year olds will be randomized into the 2 groups stratified by sex. They (parents & child) will be asked to complete a 3-day diary of food the week prior to the baseline visit and at the visit complete questionnaires (activity, eating behavior, demographics etc.). These will be used as baseline measures for all groups and for the lifestyle intervention groups to guide interventions regarding food choices and activity preferences. At the baseline visit, blood sampling, dual energy x-ray absorptiometry (DXA) and anthropometric measurements will be completed. All groups will receive simple education at the baseline visit regarding Canada's Food Guide and Canada's Activity Guide and given a 3-day diary to document their food. A registered dietitian will go through the content with them to explain how to use the guides and food-diary. Then each group will be seen at 3, 6, 9 and 12 months of study to obtain new diaries, and perform anthropometric measurements and blood biochemistry. Surveys (activity, satiety) will be taken at these visits. Body composition and bone mass will be measured at baseline, 6 and 12 months. The intervention groups will have lifestyle counseling visits at the end of months 1 through 5 to enable individualized family-child counseling (intensive phase) followed by every 3 months (establishing phase 9 months plus all receive debriefing at 12 months by a study coordinator). Intervention families will receive a monthly telephone call for any outstanding issue or to reinforce lifestyle change.

Details of Family-Child counseling at end of months 1 through 5 plus 9 mo (1.5 h visits): Intervention groups will have planning/counseling sessions for a total of 9 hours based on 5 x 1.5 h visits at the end of months 1 through 5. An additional visit at 9 mo (1.5 h) will be used to determine if new diet and activity intervention strategies are necessary over time as the child grows/matures and due to season. Counseling visits at end of months 2, 5 and 9 overlap with regular study visits and will be conducted after study data is collected to limit leading and bias (same day if need be to limit travel). All intervention planning visits will be with a registered dietitian. Both intervention groups will be instructed in detail how to use Canada's Food Guide and Activity Guide (which includes reducing screen time) and asked to set goals under the family-based behavioral intervention model of Epstein; while considering the environmental and developmental frameworks to arrive at suitable planning in the family/near environment plus suitable for the child's developmental age. The model of Epstein is grounded in the social learning theory in view of the choices, planning and reinforcement, but adapted for children/families resources and environment with reinforcement of positive behaviors. Children and families need to change together as a whole but also in support of the child being able to make decisions while away from home. This has been applied in an intervention to improve asthma control in children at and away from home.

Canada's food guide servings for Milk and Alternatives (these include for example 250 ml fluid milk, 250 ml soy beverage, 175 g yogurt, 175 kefir, 50 g cheese) is 2 per day for children 4 to 8 years of age and servings of vegetables and fruits is 5 per day. The augmented intervention group will be instructed to consume 4 servings of milk or milk products daily (these include for example 250 ml fluid milk, 175 g yogurt, 50 g cheese). The 4 servings of milk aligns with the recommended servings for 9 to 14 year old children; the age at the end of the study or soon thereafter. This intervention approach is both ethical and forward-looking. It would be unethical to counsel children and parents to not achieve the recommended 2 servings of milk and alternative products for an 8 year old. Upon completion of the study the investigators will survey families regarding sustainability of intakes at 4 servings a day - for children turning 9 years old this is the recommendation.

The intervention groups will also have counseling on other food groups to result in a healthy diet overall. Meal planning at each visit for both interventions will use Canada's Food Guide and include age appropriate serving sizes, approaches to combining foods to enhance satiety, how to incorporate snacks and fun foods, cooking methods, hidden energy, and how to specifically increase vegetables, fruit and milk intakes for the family. The examples of servings listed previously are only a few. Within each family food preferences and availability will be used to counsel towards achieving 2 or 4 servings of milk and milk products a day. Similar family-based dietary interventions have been successfully used in overweight and obese children 6 years of age and higher. The intervention groups will also actively plan to increase activity according to the Activity Guide which includes increasing activity to 90 minutes daily and decrease in non-active time by 90 minutes over 5 months (hence the visits at end of months 1 through 5). The new My Food Guide on-line at Health Canada offers a convenient tool for planning of both diet and activity that can be used over the course of the study in conjunction with the full Health Canada educational tool for planning the 5-month increase in activity and reduction in screen time. Planning with parents and children together within the context of their environment, developmental stage and food and activity preferences is anticipated to improve the program's success. A focus on fun yet feasible activities will assist both children and parents in adhering to the program. Expert researchers and health care professionals have designed both of these Health Canada tools. In fact these tools are used in the Montreal Children's Hospital obesity clinics. The activity guide has been successfully used in a 4 week family program to enhance activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 6 and 12 years of age at onset of the intervention
* Consume < 2 servings of milk and milk products but be receptive to the recommendations
* Have body mass index (BMI) over the 97 percentile for age and sex according to the World Health Organization. The Canadian Community Health Survey (CCHS)assessment of obesity used the definition by the International Obesity Task Force. This yields similar results as when using BMI percentile cut-offs proposed by the World Health Organization (WHO) for all ages of children. The WHO now has reference data available to 19 years of age. The BMI values at the 97th percentile are lower compared to the 2000 Centres for Disease Control charts (http://www.who.int/growthref/who2007_bmi_for_age/en/index.html).

Exclusion Criteria:

1. Known or suspected serious, chronic illness of childhood, such as cancer, Crohn's disease, nephrotic syndrome, rheumatic conditions, and diabetes, etc., or those with disturbances in bone, vitamin D or mineral ion metabolism including rickets, osteomalacia, liver disease, renal disease, immobilization (complete or partial), current fractures, and disorders of the parathyroid gland.
2. Use in the past 3 months, medications known to affect bone and/or mineral ion metabolism including all glucocorticoids, phosphate therapy or vitamin D analogues and any bisphosphonates.
3. Severe anemia precluding blood sampling (previously diagnosed).
4. Established diabetes mellitus (any type). Use of a glucometer and finger lance will confirm.
5. Hyperlipidemia ascribed to non-dietary causes.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Body Composition | Baseline and following 3, 6, 9 and 12 months of study participation.
  Lean mass and fat mass will be measured using a Hologic 4500A dual x-ray absorptiometry machine (DXA). For this test, children will wear standardized clothing (pyjama bottoms and T-shirt). These measures are rapid, taking a total of 5 minutes x-ray time and the low radiation (<10 uSV) will not exceed limits for x-ray exposure.

SECONDARY OUTCOMES:
Blood Biochemistry | Baseline and following 3, 6, 9 and 12 months of study participation.
  Blood samples will be drawn to examine their associations with the intervention. Analytes will include vitamin D, glucose, insulin, iron, calcium, blood lipids.
Satiety Scores | Following 12 months of study participation.
  This score will evaluate the effectiveness of the intervention on satiety. Subjects fill out a questionnaire validated in children.
Bone Mass | Baseline and following 3, 6, 9 and 12 months of study participation.
  Bone mass (whole body, lumbar spine vertebrae 1 to 4, hip bone mass and forearm) will be measured using a Hologic 4500A clinical densitometer (dual x-ray absorptiometry (DXA)). For this test, children will wear standardized clothing (pajama bottoms and T-shirt). These measures are rapid, taking a total of 5 minutes x-ray time and the low radiation (<10 uSV) will not exceed limits for x-ray exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, RD, Principal Investigator — McGill University; Celia Rodd, MD, Principal Investigator — Montreal Children's Hospital of the MUHC; Hugues Plourde, RD, PhD, Principal Investigator — McGill University
Locations (1):
- Mary Emily Clinical Nutrition Research Unit of McGill University, Sainte-Anne-de-Bellevue, Quebec, Canada

REFERENCES:
- [Derived] Cohen TR, Mak IL, Loiselle SE, Kasvis P, Hazell TJ, Vanstone CA, Rodd C, Weiler HA. Changes in Adiposity without Impacting Bone Health in Nine- to Twelve-Year-Old Children with Overweight and Obesity after a One-Year Family-Centered Lifestyle Behavior Intervention. Child Obes. 2023 Jan;19(1):46-56. doi: 10.1089/chi.2022.0008. Epub 2022 Apr 5. PMID 35384736
- [Derived] Cohen TR, Hazell TJ, Vanstone CA, Rodd C, Weiler HA. Bone Health is Maintained, While Fat Mass is Reduced in Pre-pubertal Children with Obesity Participating in a 1-Year Family-Centered Lifestyle Intervention. Calcif Tissue Int. 2017 Dec;101(6):612-622. doi: 10.1007/s00223-017-0318-8. Epub 2017 Sep 2. PMID 28866763
- [Derived] Hazell TJ, Ellery CV, Cohen TR, Vanstone CA, Rodd CJ, Weiler HA. Assessment of pedometer accuracy in capturing habitual types of physical activities in overweight and obese children. Pediatr Res. 2016 Nov;80(5):686-692. doi: 10.1038/pr.2016.133. Epub 2016 Jun 24. PMID 27486704
- [Derived] Cohen TR, Hazell TJ, Vanstone CA, Plourde H, Rodd CJ, Weiler HA. A family-centered lifestyle intervention to improve body composition and bone mass in overweight and obese children 6 through 8 years: a randomized controlled trial study protocol. BMC Public Health. 2013 Apr 25;13:383. doi: 10.1186/1471-2458-13-383. PMID 23617621